CLINICAL TRIAL: NCT05095688
Title: Relationship Between Adipose Tissue Distribution and Arterial Stiffness in Heart Failure With Preserved Ejection Fraction(HFpEF)
Brief Title: Relationship Between Adipose Tissue Distribution and Arterial Stiffness in HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2020-09-19
Record Dates: First submitted 2020-10-11; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Arterial Stiffness; Lipid Disorder
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) was considered as a heterogeneous disease with multi-organ and multi-system design, which is related to various complications, such as hypertension, obesity and arteriosclerosis. Studies have found that hypertension and obesity are respectively associated with increased arterial stiffness. However, there is still no research investigating the the relationship between lipids distribution and arterial stiffness in HFpEF patients.

DETAILED DESCRIPTION:
Before the 21st century, Heart failure with preserved ejection fraction (HFpEF) was considered as a disease with simple diastolic dysfunction, but after the 21st century, HFpEF was considered as a heterogeneous disease with multi-organ and multi-system design, which is related to various complications, such as hypertension, obesity and arteriosclerosis. Other studies have found that hypertension and obesity are respectively associated with increased arterial stiffness. However, there is still no research investigating the the relationship between lipids distribution and arterial stiffness in HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged >=18years old;
2. Diagnosed with HFpEF.

Diagnostic criteria including:

1. left ventricular ejection fraction ≥50%；
2. with the symptoms and/or signs of heart failure；
3. BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL；
4. at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction

Exclusion Criteria:

1. LVEF less than 45% at any time;
2. Severe liver failure; 3/Other causes of shortness of breath, such as severe pulmonary disease or severe chronic obstructive pulmonary disease;

4.Primary pulmonary hypertension; 5.Severe valvular disease of the left heart; 6.Chronically bedridden or incapacitated; 7.Age <18 years old.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | 1 day after admission
  The baPWV(cm/s) of HFpEF patients
adipose tissue distribution | 1 day after admission
  The visceral fat area(cm^2) in HFpEF patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No